CLINICAL TRIAL: NCT04392193
Title: Proton Particle Therapy for Cardiac Arrhythmia Extracorporeal Energy Source Ablation of Cardiac Tissue: a First Stage Early Feasibility Study
Brief Title: Proton Particle Therapy for Cardiac Arrhythmia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Konstantinos Siontis (Other)
Responsible Party: Sponsor-Investigator, Konstantinos Siontis, Principal Investigator, Mayo Clinic
Organization: Mayo Clinic (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 18-009485
Record Dates: First submitted 2020-05-14; First posted 2020-05-18 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Cardiac Arrhythmia
Keywords: Ventricular Tachycardia; Cardiac Ablation; Proton Radiation Therapy
MeSH Terms: conditions — Arrhythmias, Cardiac; Tachycardia, Ventricular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Proton Particle Therapy for Cardiac Arrhythmia (Experimental): Subjects who have an ICD with recurrent VT, VF, or VT storm who have failed one prior standard catheter-based ablation after device implantation, will subsequently undergo particle-based extracorporeal ablation.
  Interventions: Radiation: Proton Particle Therapy

INTERVENTIONS:
Radiation: Proton Particle Therapy — Proton therapy will be delivered in a single fraction using the Probeat-V system

SUMMARY:
Researchers are gathering information on the safety and effectiveness of proton radiation therapy in reducing the number of ventricular tachycardia (VT) episodes in subjects who continue to experience VT despite treatment with an implantable cardioverter defibrillator (ICD) and undergoing a previous catheter ablation.

DETAILED DESCRIPTION:
Proton therapy has been approved by the U.S. Food and Drug Administration (FDA) for cancer patients, including tumors in the heart, but not for treating heart rhythm disorders. The use of proton radiation therapy to treat heart rhythm disorders including VT and ventricular fibrillation (VF) is new and investigational; however, the FDA has approved proton therapy to treat abnormal rhythm disorders for this study. The development of a proton radiation therapy approach could be of substantial value in providing alternative therapy to either drug therapy or catheter-based ablation. With appropriate development, this therapy may be successful in the primary or secondary elimination of arrhythmias.

Participants will be followed at 1 and 2 weeks, 1, 3, 6, 12 and 24-month intervals following treatment throughout the trial.

Participant involvement will last approximately two years from the time of the proton radiation therapy procedure or until the last subject enrolled completes a 24 month follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Prior myocardial infarction, or non-ischemic disease, resulting in myocardial dysfunction
2. EF <50%
3. An implanted ICD device as secondary prevention for monomorphic VT/VF (MMVT/MMVF). This includes patients who receive a device for primary prevention and then have recurrent sustained monomorphic VT or VF.
4. Have failed a prior catheter-based ablation for VT/VF after device implantation or have a contraindication to repeat ablation and have failed reasonable drug options over the 9 months prior to consideration of particle therapy.
5. Repeat ablation from an epicardial venue in the absence of prior cardiac surgery, or where such an ablation is felt to be inappropriate in the view of the PI.
6. Electrocardiographic documentation of 2 additional episodes of recurrent, sustained monomorphic ventricular tachycardia (MMVT) and/or PVC induced VT or VF that are terminated by ATP or ICD shocks (by device interrogation) over the past 9 months, since the sentinel ablation (see criteria #4). Also included, incessant VT that does not fall within device parameters for activation of ATP or shock delivery or is refractory to medication titration.
7. Age <=80 years.

Exclusion Criteria:

1. VT in the absence of cardiomyopathy.
2. Reversible causes of VT including thyroid disorders, acute alcohol intoxication, recent major surgical procedures, trauma, or VT clearly produced by recurrent ischemia.
3. Multiple (e.g.>3) clinical VT morphologies that are thought to originate from widely disparate RV or LV areas.
4. Recent cardiac events including MI, PCI, or valve or bypass surgery in the preceding 3 months, or anticipated in the next 3 months.
5. Hypertrophic obstructive cardiomyopathy (HOCM) >Class IV
6. Progressive Class IV angina, or Class IV CHF (including past, or planned heart transplantation).
7. Heritable arrhythmias or increased risk for torsade de pointes with Class I or III drugs.
8. Prior surgical interventions for VT such as an encircling ventriculotomy procedure.
9. Contraindication to appropriate anti-coagulation therapy after ablation.
10. Renal failure requiring dialysis.
11. Prior therapeutic radiation therapy to the left chest that would preclude safe ablation of the cardiac target in the judgement of the radiation oncologist.
12. Medical conditions limiting expected survival <1 year.
13. Women of child bearing potential (unless post-menopausal or surgically sterile)
14. Participation in any other clinical mortality trial (participation in other non-mortality trials should be reviewed with the clinical trial management center)
15. Unable to give informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2021-03-19 (Actual); Primary Completion 2024-03-09 (Actual); Study Completion 2024-03-09 (Actual)

PRIMARY OUTCOMES:
Mortality | 2 years
  Total number of subject deaths
Implantable Cardioverter Defibrillator (ICD) Shocks | 2 years
  Total number of recurrent ICD shocks
Recurrent Ventricular Tachycardia (VT) | 2 years
  Total number of recurrent VT requiring repetitive antitachycardia pacing (ATP) device therapy
Cardiac Arrest | 2 years
  Total number of cardiac arrests

CONTACTS AND LOCATIONS:
Overall Officials: Konstantinos Siontis, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No